CLINICAL TRIAL: NCT02698761
Title: A Comprehensive Care Plan for Pediatric Patients With Vaso-Occlusive Crises
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Standard of care changed
Sponsor: Valley Anesthesiology Consultants (Other)
Collaborators: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15-129
Record Dates: First submitted 2016-02-01; First posted 2016-03-04 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Sickle Cell Disease; Sickle Cell Crisis; Vaso-Occlusive Crises
Keywords: Vaso-Occlusive Crises; Sickle Cell Disease; Decreasing Length of Stay; Comprehensive Care Plan
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Patient will receive standard of care. Subject will have an actiwatch to compare activity and sleep habits. Nursing staff will be aware of study presence but will not receive any specific instruction for the patient.
- Comprehensive Care Plan (Experimental): Patient will abide by the comprehensive care plan and sign an agreement stating compliance. Subject will have an actiwatch to compare activity and sleep habits. Nursing staff will be notified of study and support patient's compliance with study procedures.
  Interventions: Other: Comprehensive Care Plan

INTERVENTIONS:
Other: Comprehensive Care Plan — Care Plan
  1. Patient Controlled Analgesia (PCA). PCA will be initiated and managed at the discretion of the Pain Management team.
  2. Other Medications. All medications will be given during daytime hours, if possible.
  3. Pain Psychology.
  4. Physical Therapy. Patient is expected to spend time out of bed by Day 2 participating in light activity.
  5. Sleep Hygiene. Patient sleeps between the hours of 10 PM and 5 AM daily. Window blinds open by 8 AM. Patient must be awake and ready to participate in therapy by 9 AM.
  6. Extracurricular. TV, phone, computer, and video games only between hours of 4-9 PM (computer okay outside of hours only for school work).
  7. Other. Patient will eat meals during regular daytime hours (e.g. breakfast consumed before 9 am) and shower daily.
  Arms: Comprehensive Care Plan

SUMMARY:
Sickle cell disease (SCD) is the most common inherited blood disorder affecting 80,000 to 90,000 individuals in the United States.[10] There are 13,000 hospital admissions for a sickle cell crises, costing $448 million dollars annually.[10] In our hospital, the sickle cell population is known to have some of the longest length of stays. Between October 2014 and September 2015, there were 89 admissions for a vaso-occlusive crisis with an average length of stay of 6 days and 12 admissions greater than 10 days and 5 admissions greater than 20 days.

We propose to evaluate the feasibility of the new CPP in a pilot randomized control trial to determine if pain and length of stay can be reduced in patients with sickle cell disease. We also propose to evaluate a sleep regimen to determine if this can reduce the hospital stay and help with pain. We hypothesize increased physical activity and proper sleep, as implemented in the CPP, are correlated with decreased hospital length of stay and decreased pain. Additionally, we believe that creating a standardized nighttime environment at the hospital will help the children stay in their circadian rhythm thus promoting improved sleep and a more effective inpatient disease management.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) disease is inherited as an autosomal recessive trait that results in several interactive processes: polymerization of hemoglobin S (HbS), hemolysis, nitric oxide depletion, and vaso-occlusion.[3] The most common manifestations of sickle cell disease are vaso-occlusive pain events, specifically dactylitis which typically occurs as the first clinical manifestation.[4] As patients age, the early onset peripheral pain moves to more central regions resulting in increased severity of vaso-occlusive crises.[4] Pain from the blockage of sickeled cells in vessels causes poor blood flow to a localized area. There are few clinical and laboratory findings to indicate the severity of pain associated with sickle cell crisis,[4] making it difficult for a physician to identify the amount of pain the patient actually experiences. Length of stay in the hospital depends largely on physician discretion and patient report.

Sleep is instrumental to many aspects of physical and emotional health during childhood and adolescence. Sleep disruption from pain is a significant concern in patients with sickle cell disease due to the prevalence of their acute and chronic pain.[7] In a study conducted by Daniel et al., sickle cell patients between 4-10 years old, were more likely to exhibit disrupted sleep, specifically night-waking and sleep-disordered breathing, than children who were not diagnosed with sickle cell disease from similar demographic backgrounds. [7] Furthermore, children with more severe forms of sickle cell disease were reported to have more restless sleep than children with less severe forms. [7] Overall, the literature suggests that sleep disruptions may interfere with children's daily functions, along with their ability to cope with SCD and its complications.[7] Daniel et al. recommends discussing ways to improve sleep habits with children suffering from SCD because it may increase efficacy in pain management, priapism, and enuresis.[7] Another study by Valrie etal., suggests that poor quality of sleep is correlated with increased occurrence of sickle cell disease pain the following day.[9] They also discovered that high pain severity was related to poor sleep quality and this relationship was exacerbated during stressful situations.[9] Developing a suitable sleeping environment (e.g. removing the television, or limiting the lighting) will maximize sleep efficacy resulting in better health outcomes and quality of life.[7] There has been minimal research on evaluating the relationship between exercise and sickle cell disease in children and adolescents. Studies conducted on sickle cell disease in adults with respect to the effects of exercise have produced mixed results partly due to patient comorbid illnesses. In 2012, Chirico et al. compared two fitness level group including, subjects who did not partake in regular physical activity for two years prior to the study versus subjects who partook in regular, weekly physical activity for several years leading up to the study. [5] Both groups contained sickle cell trait carriers and subjects with normal hemoglobin. [5] Subjects performed an incremental maximum exercise test while data was collected on heart rate via a chest monitor and on oxidative stress levels via blood samples at various points following completion of the exercise task. [5] Results indicated regular physical activity helped to blunt the increase in oxidative stress and the decrease in nitric oxide metabolism and up regulation of antioxidant enzyme activities in response to exercise in sickle cell trait carriers. [5] These findings suggest an attenuated sickle cell crisis in the subjects with regular exercise when compared with the sedentary group.

Presently, at Phoenix Children's Hospital, no protocol exists for management of sleep and exercise in sickle cell patients. The most relevant policy named "Parenting and Visitation" includes guidelines regarding sleep and visiting hours but these are not well enforced. In our hospital, the sickle cell population is known to have some of the longest length of stays. Between October 2014 and September 2015, there were 89 admissions for a vaso-occlusive crisis with an average length of stay of 6 days and 12 admissions greater than 10 days and 5 admissions greater than 20 days. Prior research suggests that implementation of standardized care (e.g. order sets, protocols, and flowcharts) can improve compliance and patient outcomes [8], reduce overall length of stay, and mitigate costs. Therefore, we have developed a new comprehensive care plan (CPP) that enhances standard of care by including the following care aspects:

1. Patient Controlled Analgesia (PCA). PCA will be initiated and managed at the discretion of the Pain Management team. Naloxone infusion will be available for opioid related side effects. Once tapered, patients will be transitioned to oral opioids to be administered as needed. Patients will be discharged home, when appropriate, with oral opioids and weaning instructions.
2. Other Medications. All medications will be given during daytime hours, if possible. All home medications will be continued while inpatient. Ketorolac will be given intravenously every 6 hours for 12 doses then switched to ibuprofen by mouth every 6 hours until discharge home. Stool softeners will be utilized while on narcotics to prevent constipation. A clonidine patch may be used for adjunct analgesia and anxiolysis. A lidocaine patch may be used for localized pain.
3. Pain Psychology. Consultations will begin on Day 2 and continue as needed. The psychologist will teach the patient sleep hygiene techniques, and non-pharmacologic pain management skills including: distraction, diaphragmatic breathing, progressive muscle relaxation, and guided imagery with medical hypnosis.
4. Physical Therapy. Consultations will begin on Day 2 and continue as needed. Patient is expected to spend time out of bed by Day 2 participating in light activity.
5. Sleep Hygiene. Will be introduced to the experimental group. Patient must sleep between the hours of 10 PM and 5 AM daily. Window blinds will be open by 8 AM. Patient must be awake and ready to participate in therapies by 9 AM. Napping will be at the discretion of the physician. Practitioners should examine care orders critically, such as routine vital signs, and determine if it is safe and/or appropriate to defer these during sleep. Room lights will be turned off to help promote the circadian rhythm. No video games, television, cell phones, or computers will be allowed during this time.
6. Extracurricular. Will participate in child life activities as recommended (e.g. Playroom, or Zone). TV, phone, computer, and video games only between hours of 4-9 PM (computer okay outside of hours only for school work).
7. Other. Patient will eat meals during regular daytime hours (e.g. breakfast consumed before 9 am) and shower daily. No overnight visitors will be allowed.

We propose to evaluate the feasibility of the new CPP in a pilot randomized control trial to determine if pain and length of stay can be reduced in patients with sickle cell disease. We also propose to evaluate a sleep regimen to determine if this can reduce the hospital stay and help with pain. We hypothesize increased physical activity and proper sleep, as implemented in the CPP, are correlated with decreased hospital length of stay and decreased pain. Additionally, we believe that creating a standardized nighttime environment at the hospital will help the children stay in their circadian rhythm thus promoting improved sleep and a more effective inpatient disease management.

Specific Aims Primary: To determine the feasibility and efficacy of the CPP to reduce pain and length of stay in patients with sickle cell disease.

A.To evaluate if patients who follow the CPP physical activity regimen will have less pain and shorter hospital stay than patients receiving standard of care.

B.To measure if patients who follow the CPP sleep activity regimen will have less pain and shorter hospital stay than patients receiving standard of care.

Study Design This is a prospective pilot study of 20 subjects who have sickle-cell disease and are admitted to Phoenix Children's Hospital for an acute vaso-occlusive crisis. Patients will be randomized via a random number generator with equal probability of assignment to either CPP (experimental) or standard of care (control) trial arm. Eligible subjects and their family will be approached during the first day of hospital admission for consent to participate and randomization. After randomization, all subjects will be given multiple questionnaires to evaluate their current sleep habits, activity levels, and psychological constructs Procedures During the enrollment visit, questionnaires will be administered to every subject to evaluate current sleep habits, activity levels, pain, and quality of life. Subjects will receive the Actiwatch Spectrum Pro and be given instructions on how to use it.

Control Group: Patient will receive standard of care. Nursing staff will be aware of study presence but will not receive any specific instruction for the patient.

Experimental Group: During the enrollment visit, patient will go over the new comprehensive care protocol with the study staff and will sign the agreement stating compliance. Patient will be given a copy of the comprehensive care plan for reference. Nursing staff will be aware of study's presence and will help to support patient's compliance with sleep and other procedures according to care plan.

Discharge Study staff will closely follow the patient's progress in the hospital. Once patient is ready for discharge, they will have a visit with study investigators and be given one final PedsQL™ to complete. An additional questionnaire will be given to the experimental group asking their opinion about the CPP. The Actiwatch Spectrum Pro will be collected from the patients and be properly disinfected.

Measurement/Assessments Actiwatch Spectrum Pro Monitoring Device The Actiwatch Spectrum Pro activity device will continuously monitor activity (active minutes), sleep (minutes slept and quality) and allow the subject to input their numerical pain or fatigue rating. At the end of the patient's trial, the data will be extracted from the actiwatch and placed into the patient's alphanumeric account that is monitored by the research personnel. Patients or families will not have access to the accounts. We will examine the minutes of activity per day and minutes of sleep per day and compare it to the pain scores recorded by looking at the data extracted from the Actiwatch Spectrum Pro.

Analysis Baseline characteristics will be summarized within the two care groups using descriptive statistics including count and percent for categorical variables and the mean and standard deviation (median and interquartile ranges) for continuous variables. Evaluation of the CPP with length of stay will be done using the T-test or the Kruskal-Wallis test, depending on the length of stay distribution. Analysis of variance for repeated measures will assess the effect of time on pain scores within care groups. Differences in mean cumulative pain scores between care groups will also be examined daily during hospital stay.

Additional analyses will investigate the association of care components, physical activity and sleep, with length of stay and pain scores using appropriate statistical methods as described above. All statistical tests will have a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Children between 12 and 18 years of age who are admitted to the hospital for an acute vaso-occlusive crisis
* Patients must require a demand PCA and able to tolerate oral pain medications

Exclusion Criteria:

* - Requires a continuous PCA
* Unwilling to be compliant with the assigned arm of study (e.g. Non-compliance with sleep or visiting regimen, or questionnaires)
* Non-English speaking child or parent (questionnaires not available/validated in another language)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Length of Stay | 2 Years
  Length of Stay in Days

SECONDARY OUTCOMES:
Pain Scores | 2 Years
  pain scores assessed daily for each patient using the (Visual Analog Scale) VAS scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morrissey LK, Shea JO, Kalish LA, Weiner DL, Branowicki P, Heeney MM. Clinical practice guideline improves the treatment of sickle cell disease vasoocclusive pain. Pediatr Blood Cancer. 2009 Mar;52(3):369-72. doi: 10.1002/pbc.21847. PMID 19023890
- [Background] Vijenthira A, Stinson J, Friedman J, Palozzi L, Taddio A, Scolnik D, Victor C, Kirby-Allen M, Campbell F. Benchmarking pain outcomes for children with sickle cell disease hospitalized in a tertiary referral pediatric hospital. Pain Res Manag. 2012 Jul-Aug;17(4):291-6. doi: 10.1155/2012/614819. PMID 22891195
- [Background] Chirico EN, Martin C, Faes C, Feasson L, Oyono-Enguelle S, Aufradet E, Dubouchaud H, Francina A, Canet-Soulas E, Thiriet P, Messonnier L, Pialoux V. Exercise training blunts oxidative stress in sickle cell trait carriers. J Appl Physiol (1985). 2012 May;112(9):1445-53. doi: 10.1152/japplphysiol.01452.2011. Epub 2012 Feb 9. PMID 22323645
- [Background] Fonarow GC, Gawlinski A, Moughrabi S, Tillisch JH. Improved treatment of coronary heart disease by implementation of a Cardiac Hospitalization Atherosclerosis Management Program (CHAMP). Am J Cardiol. 2001 Apr 1;87(7):819-22. doi: 10.1016/s0002-9149(00)01519-8. PMID 11274933